CLINICAL TRIAL: NCT03256344
Title: A Phase 1b Study of Talimogene Laherparepvec in Combination With Atezolizumab in Subjects With Triple Negative Breast Cancer and Colorectal Cancer With Liver Metastases
Brief Title: Study of Talimogene Laherparepvec With Atezolizumab for Triple Negative Breast Cancer and Colorectal Cancer With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20140299
Record Dates: First submitted 2017-08-08; First posted 2017-08-22 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Triple Negative Breast Cancer; Metastatic Colorectal Cancer
Keywords: Liver Metastases
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Colorectal Neoplasms | interventions — talimogene laherparepvec; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Talimogene Laherparepvec with Atezolizumab: Triple Negative Breast Cancer (TNBC) (Experimental): Participants with TNBC with liver metastases administered intrahepatic injection of talimogene laherparepvec into liver metastases via guided injection (either ultrasound or computerized tomography) on Day 1 of each cycle for a maximum of 12 cycles, where each cycle is 21 days. Participants administered 10^6 plaque-forming units/milliliter (PFU/mL) on Day 1 of Cycle 1 and 10^8 PFU/mL on Day 1 of each cycle thereafter. Participants also administered 1200 mg atezolizumab via intravenous injection on Day 1 of each cycle.
  Interventions: Biological: Talimogene Laherparepvec; Biological: Atezolizumab
- Talimogene Laherparepvec with Atezolizumab: Colorectal Cancer (CRC) (Experimental): Participants with CRC with liver metastases administered intrahepatic injection of talimogene laherparepvec into liver metastases via guided injection (either ultrasound or computerized tomography) on Day 1 of each cycle for a maximum of 12 cycles, where each cycle is 21 days. Participants administered 10^6 PFU/mL on Day 1 of Cycle 1 and 10^8 PFU/mL on Day 1 of each cycle thereafter. Participants also administered 1200 mg atezolizumab via intravenous injection on Day 1 of each cycle.
  Interventions: Biological: Talimogene Laherparepvec; Biological: Atezolizumab

INTERVENTIONS:
Biological: Talimogene Laherparepvec — Virally based anti-cancer immunotherapy given by direct injection into tumors.
  Other Names: IMLYGIC
Biological: Atezolizumab — A monoclonal antibody given by intravenous injection.
  Other Names: MPDL3280A

SUMMARY:
Approximately 36 DLT-evaluable subjects will be enrolled in this study. The locations of the study will be in the United States, Australia, Europe and Switzerland.

The goal of this study is to evaluate the safety of intrahepatic injection (directly into the liver) of talimogene laherparepvec in combination with intravenously administered atezolizumab in subjects with triple negative breast cancer and colorectal cancer with liver metastases.

DETAILED DESCRIPTION:
The Screening period is 28 days prior to study enrollment. This study has 2 Cohorts. Cohort 1: Triple Negative Breast Cancer and Cohort 2: Colorectal Cancer. These cohorts will enroll in parallel. There will be a Safety Follow-up period and a Long Term Follow-up period.

Drug Administration: The participants will receive the study drugs in cycles. If the participants are found to be eligible to take part in this study, they will receive talimogene laherparepvec as an injection into the hepatic (liver) metastatic sites on Day 1 of each cycle along with receiving atezolizumab by intravenous infusion on Day 1 of each cycle. Each cycle is 21 days for 6 cycles. There is an option for an additional 6 cycles after the first 6 intra-hepatic cycles. After the first radiographic assessment at week 10, if all injectable liver lesions have been injected but the 4.0 mL maximum volume has not been used, injection of clinically assessed non-hepatic cutaneous, subcutaneous, and nodal tumor lesions with or without ultrasound guidance will be permitted. Liver lesions should be prioritized over cutaneous, subcutaneous and nodal lesions.

Treatment will continue until a participant experiences a DLT (Dose Limiting Toxicity) evaluated in the DLT period (which is 2 cycles from initial dose), has CR (Complete Response), has need for an alternative anticancer therapy or experiences a safety concern.

Study Visits: Cycle 1 to Cycle 12 - The participant will have a physical exam along with vital signs and ECOG (Eastern Cooperative Oncology Group) performance level assessment. Blood (about 2 Tablespoons) will be drawn for routine tests and to check the immune system. Adverse events and medications taken will be reviewed on each cycle.Biomarkers will be taken on cycles 1, 2, 3, 6, and safety FU. Tumor Markers (special lab tests associated with the cancer, such as particular proteins) will be completed will be take on cycles 1, 4, 7, 10, 13, every 3 cycles and SFU.

Central lab tests will be completed on cycles 1, 2, 3, and 6 and safety FU. Cycle 1 Archived (prior stored) tumor sample will be obtained. Also, a liver tumor biopsy will be completed at Cycles 1, 3 and 6.

Response Assessments will be completed at Screening and again at Cycles 4, 7, 10, 13 and every 3 cycles.

Throughout the trial a swab for Herpetic tumor will be obtained within 3 days of the event.

Cycle 1 to 12- The exposure to talimogene laherparepvec by the subject's healthcare provider and household member caregiver will be reviewed. Cycles 1, 3, 6-Liver tumor biopsy will be completed. Cycles 4, 7, 10, 13 and every 3 cycles -Response assessments will be completed by radiographic and clinical tumor assessment.

Length of Treatment:

A maximum for 12 cycles of talimogene laherparepvec are allowed during the study. The participant may continue taking the study drug for as long as the doctor thinks it is in their best interest. The participant will no longer be able to take the study drug if the disease gets worse, or if they are unable to follow study directions.

Safety Follow-up Visit:

Safety Follow-up visit will be performed about 30 days after the last dose of study treatment.

The participant will have a physical exam, have vital signs taken, assessment of ECOG status and have weight measured. Adverse events will be assessed as well as the concominant medications. Routine bloodwork and tumor markers will be taken.

Exposure to talimogene laherparepvec by the healthcare providers of the participant and/or close contacts will be assessed.

Long-Term Follow-up Visits: Participants will be followed for survival every 12 weeks from the date of the safety follow-up visit until approximately 24 months after the last subject is enrolled. Subsequent cancer treatments will be collected as part of the long-term follow-up survival assessment. This is an investigational study. The study doctor can explain how the study drugs are designed to work.

ELIGIBILITY:
Inclusion Criteria:

* Criteria1, Participant provided informed consent prior to any study-specific activities/procedures.
* Criteria 2, Confirmation of triple negative breast cancer or colorectal cancer with liver metastases by laboratory testing.
* Criteria 3, Subjects with triple negative breast cancer with liver metastases, or subjects with colorectal cancer with liver metastases are eligible if they have had disease progression during or after one or more prior standard of care systemic anti-cancer therapy (eg,chemotherapy, targeted therapy) for metastatic disease or if they progress during or within 6 months of receiving adjuvant therapy. If subjects, in the opinion of the investigator, are deemed not appropriate candidates for systemic anti-cancer therapy for metastatic disease or if they refuse systemic anti-cancer therapy for metastatic disease, they may be eligible after investigator discussion with Sponsor medical monitor for approval.
* Criteria 4, Participants have measurable disease which is equal to one or more metastatic liver lesions that can be accurately and serially measured that are greater than or equal to 1 cm dimension and for which the longest diameter is greater or equal to 1 cm as measured by CT (Computed Tomography) scan or magnetic resonance imaging. The metastatic liver lesion(s) must not be in an area that received prior localized therapies.
* Criteria 5, Metastatic liver lesions for injection must be without necrosis (dead tissue )and must be be located where any tumor swelling will not lead to gall bladder tract obstruction or lead to bleeding risk.
* Criteria 6, Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* Criteria 7, Life expectancy greater than or equal to 5 months.
* Criteria 8, Adequate organ function within 4 weeks prior to enrollment. This includes hematology, renal, hepatic and blood-clotting functions as defined by protocol.
* Criteria 9, Female subjects of childbearing potential should have a negative serum pregnancy test within 1 week prior to enrollment.
* Criteria 10, Other Inclusion Criteria May Apply.

Exclusion criteria:

* Criteria 1, Participant is a candidate for hepatic surgery or local regional therapy of liver metastases with curative intent.
* Criteria 2, More than one third of the liver is estimated to be involved with metastases.
* Criteria 3, There is invasion by cancer into the main blood vessels such as the portal vein, hepatic vein or the vena cava.
* Criteria 4, Participant is currently receiving or has received liver metastatic-directed therapy ( eg: radiation, ablation, embolization) less than 4 wks prior to enrollment or hepatic surgery.
* Criteria 5, History of other malignancy within the past 5 years prior to enrollment with some exceptions, as outlined in the protocol.
* Criteria 6, Active or untreated central nervous system (CNS) metastases per CT or magnetic resonance imagine (MRI) evaluation during screening.
* Participants with a history of CNS metastases are eligible provided they are stable and meet the criteria details in the protocol.
* Criteria 7, Other Medical Conditions as noted in the protocol.
* Criteria 8, Other Exclusion Criteria May Apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - Columbia University Medical Center, New York, New York
  - Stony Brook University, Stony Brook, New York
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Breast Cancer Research Centre - WA, Nedlands, Western Australia
- Belgium (2):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Germany (3):
  - Charite UniversitÃ¤tsmedizin Berlin, CharitÃ© Campus Virchow-Klinikum, Berlin
  - UniversitÃ¤tsklinikum Bonn, Bonn
  - UniversitÃ¤tsklinik TÃ¼bingen, TÃ¼bingen
- Spain (3):
  - Hospital del Mar, Barcelona, CataluÃ±a
  - Hospital General Universitario Gregorio MaraÃ±on, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
- Switzerland (2):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Hecht JR, Raman SS, Chan A, Kalinsky K, Baurain JF, Jimenez MM, Garcia MM, Berger MD, Lauer UM, Khattak A, Carrato A, Zhang Y, Liu K, Cha E, Keegan A, Bhatta S, Strassburg CP, Roohullah A. Phase Ib study of talimogene laherparepvec in combination with atezolizumab in patients with triple negative breast cancer and colorectal cancer with liver metastases. ESMO Open. 2023 Apr;8(2):100884. doi: 10.1016/j.esmoop.2023.100884. Epub 2023 Feb 28. PMID 36863095
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 15 research centers in Australia, Belgium, Germany, Spain, Switzerland and the United States.
Pre-assignment Details: Participants were enrolled between 19 March 2018 and 03 December 2021. A total of 11 subjects with triple negative breast cancer were enrolled and 25 subjects with colorectal cancer.
Groups:
- Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC): Participants with TNBC with liver metastases were administered intrahepatic injection of talimogene laherparepvec into liver metastases via guided injection (either ultrasound or computerized tomography) on Day 1 of each cycle for a maximum of 12 cycles, where each cycle was 21 days. Participants were administered 10^6 plaque-forming units/milliliter (PFU/mL) on Day 1 of Cycle 1 and 10^8 PFU/mL on Day 1 of each cycle thereafter. Participants were also administered 1200 mg atezolizumab via intravenous injection on Day 1 of each cycle.
- Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC): Participants with CRC with liver metastases were administered intrahepatic injection of talimogene laherparepvec into liver metastases via guided injection (either ultrasound or computerized tomography) on Day 1 of each cycle for a maximum of 12 cycles, where each cycle was 21 days. Participants were administered 10^6 PFU/mL on Day 1 of Cycle 1 and 10^8 PFU/mL on Day 1 of each cycle thereafter. Participants were also administered 1200 mg atezolizumab via intravenous injection on Day 1 of each cycle.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Started | 11 | 25
Received Talimogene Laherparepvec | 8 | 23
Received Atezolizumab | 10 | 24
Safety Analysis Set (All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.) | 10 | 24
Completed | 1 | 0
Not Completed | 10 | 25
Not completed — Death | 6 | 22
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC) | Total
Number analyzed (Participants) | 11 | 25 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 25
  >=65 years | 1 | 10 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 13 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 24 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 10 | 22 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: Toxicities were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A DLT was considered as any of the below, if judged by the investigator to be related to either treatment:
  * Grade ≥ 4 neutropenia (absolute neutrophil count [ANC] < 500/μl) lasting ≥ 7 days
  * Grade ≥ 3 febrile neutropenia
  * Grade ≥ 4 thrombocytopenia
  * Grade ≥ 4 anemia
  * Grade ≥ 4 rash
  * Serious herpetic events
  * Grade ≥ 3 symptomatic hepatic toxicities that do not resolve to Grade ≤ 2 within 48 hours or Grade ≥ 3 asymptomatic hepatic toxicities that do not resolve to Grade ≤ 1 within 3 weeks of onset
  * Grade ≥ 3 non-hematologic, non-hepatic organ toxicity
  * Grade 5 toxicity (ie, death)
  * Any other intolerable toxicity leading to permanent discontinuation of treatment
  DLTs were to occur within the DLT evaluation period, defined as the period between the initial 10^6 PFU/mL dose and 3 weeks following the initial 10^8 PFU/mL dose or the start of Cycle 3, whichever occurred first.
Time Frame: From Day 1 up to the start of Cycle 3 (each cycle is 21 days)
Population: DLT Analysis Set: All participants who had opportunity to receive treatment for 2 cycles from the time of initial dose of study treatment and who had received 2 doses of talimogene laherparepvec and 2 doses of atezolizumab in combination or had a DLT during the DLT-evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 5 | 18
Participants | 0 | 3

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the incidence rate of either a complete response (CR) or partial response (PR) based on modified immune-related response criteria simulating Response Evaluation Criteria in Solid Tumors(irRC-RECIST) criteria. A CR was a complete disappearance of all lesions and a PR was a decrease in tumor burden 30% or more relative to baseline.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Percentage of Participants | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 14.2]

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was defined as the best visit response based on modified irRC-RECIST criteria:
  * CR: a complete disappearance of all lesions
  * PR: a decrease in tumor burden 30% or more relative to baseline
  * Stable disease (SD): neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for progressive disease (PD)
  * PD: an increase in tumor burden of 20% or more and at least 5 mm absolute increase relative to nadir (minimum recorded tumor burden)
  * Unevaluable (UE): any lesion present at baseline which was not assessed or was unable to be evaluated leading to an inability to determine the status of that particular tumor
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Participants
  CR | 0 | 0
  PR | 1 | 0
  SD | 1 | 1
  PD | 3 | 4
  UE | 3 | 14
  Not done | 2 | 5

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of an initial response that is subsequently confirmed to the earlier of PD per modified irRC RECIST or death. Participants who have not ended their response at the time of analysis were censored at the last evaluable tumor assessment.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Responders in Safety Analysis Set: All participants in safety analysis set who received at least 1 dose of talimogene laherparepvec or atezolizumab who had a best overall response of CR/PR at the time of analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 1 | 0
Months | NA [NA to NA] — Not calculable as only 1 participant achieved response. |

5. Secondary Outcome: Lesion Level Response in Injected Tumor Lesions
Description: Responses for individual tumor lesions for hepatic and non-hepatic tumors injected wtih treatment were assessed for the following responses:
  * Lesion complete response rate (L-CRR): Disappearance of lesion
  * Lesion partial response rate (L-PRR): Decrease in tumor burden 30% or more relative to baseline
  * Lesion objective response rate (L-ORR): Either a L-CRR or L-PRR based on modified irRC-RECIST criteria
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Injected Lesion Analysis Set: Any target lesion and new measurable lesion that was injected from the participants who had received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 8 | 20
Number analyzed (Lesions) | 13 | 28
Lesions
  L-CRR - Hepatic | 0 [0.0 to 24.7] | 0 [0.0 to 12.3]
  L-CRR - Non-hepatic: number analyzed (Participants) | 0 | 0
  L-CRR - Non-hepatic: number analyzed (Lesions) | 0 | 0
  L-CRR - Overall | 0 [0.0 to 24.7] | 0 [0.0 to 12.3]
  L-PRR - Hepatic | 1 [0.2 to 36.0] | 0 [0.0 to 12.3]
  L-PRR - Non-hepatic: number analyzed (Participants) | 0 | 0
  L-PRR - Non-hepatic: number analyzed (Lesions) | 0 | 0
  L-PRR - Overall | 1 [0.2 to 36.0] | 0 [0.0 to 12.3]
  L-ORR - Hepatic | 1 [0.2 to 36.0] | 0 [0.0 to 12.3]
  L-ORR - Non-hepatic: number analyzed (Participants) | 0 | 0
  L-ORR - Non-hepatic: number analyzed (Lesions) | 0 | 0
  L-ORR - Overall | 1 [0.2 to 36.0] | 0 [0.0 to 12.3]

6. Secondary Outcome: Lesion Level Response in Uninjected Tumor Lesions
Description: Responses for individual tumor lesions for hepatic and non-hepatic tumors that were not injected with treatment were assessed for the following responses:
  * L-CRR: Disappearance of lesion
  * L-PRR: Decrease in tumor burden 30% or more relative to baseline
  * L-ORR: Either a L-CRR or L-PRR based on modified irRC-RECIST criteria
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Uninjected Lesion Analysis Set: Any target lesion and new measurable lesion that was never injected from the participants who had received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 22
Number analyzed (Lesions) | 24 | 94
Lesions
  L-CRR - Hepatic: number analyzed (Lesions) | 15 | 50
  L-CRR - Hepatic | 0 [0.0 to 21.8] | 0 [0.0 to 7.1]
  L-CRR - Non-hepatic: number analyzed (Lesions) | 9 | 44
  L-CRR - Non-hepatic | 0 [0.0 to 33.6] | 0 [0.0 to 8.0]
  L-CRR - Overall | 0 [0.0 to 14.2] | 0 [0.0 to 3.8]
  L-PRR - Hepatic: number analyzed (Lesions) | 15 | 50
  L-PRR - Hepatic | 0 [0.0 to 21.8] | 1 [0.1 to 10.6]
  L-PRR - Non-hepatic: number analyzed (Lesions) | 9 | 44
  L-PRR - Non-hepatic | 1 [0.3 to 48.2] | 0 [0.0 to 8.0]
  L-PRR - Overall | 1 [0.1 to 21.1] | 1 [0.0 to 5.8]
  L-ORR - Hepatic: number analyzed (Lesions) | 15 | 50
  L-ORR - Hepatic | 0 [0.0 to 21.8] | 1 [0.1 to 10.6]
  L-ORR - Non-hepatic: number analyzed (Lesions) | 9 | 44
  L-ORR - Non-hepatic | 1 [0.3 to 48.2] | 0 [0.0 to 8.0]
  L-ORR - Overall | 1 [0.1 to 21.1] | 1 [0.0 to 5.8]

7. Secondary Outcome: Durable Response Rate (DRR)
Description: DRR was defined as the percentage of participants with an objective response with a DOR of at least 6 months.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Percentage of Participants | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 14.2]

8. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants that have a best overall response in one of the following categories: CR/PR/SD.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Percentage of Participants | 20.0 [2.5 to 55.6] | 4.2 [0.1 to 21.1]

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from first dose to the date of first of confirmed disease progression per modified irRC-RECIST criteria, or death (whichever occurred first). Results were estimated using the Kaplan-Meier method.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Months | 5.4 [1.0 to NA] — Upper limit was not estimable. | 3.1 [2.1 to 5.2]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death from any cause. Results were estimated using the Kaplan-Meier method.
Time Frame: Every 12 weeks (± 28 days) up to approximately 3.5 years.
Population: Safety Analysis Set: All participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
Number analyzed (Participants) | 10 | 24
Months | 19.2 [1.5 to NA] — Upper limit was not estimable. | 4.0 [2.8 to 6.6]

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 3.5 years.
Description: All-Cause Mortality is reported for all enrolled participants. Serious and Other Adverse Events are reported for the Safety Analysis Set defined as all participants who received at least 1 dose of talimogene laherparepvec or atezolizumab.
Arm/Group | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC)
All-Cause Mortality (participants affected / at risk) | 6/11 | 22/25
Serious Adverse Events (participants affected / at risk) | 4/10 | 12/24
Other Adverse Events (participants affected / at risk) | 8/10 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) (N=10) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC) (N=24)
Cardiac failure (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour hyperprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec With Atezolizumab: Triple Negative Breast Cancer (TNBC) (N=10) | Talimogene Laherparepvec With Atezolizumab: Colorectal Cancer (CRC) (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 5
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 8
Asthenia (General disorders) | 0 | 4
Chills (General disorders) | 4 | 2
Fatigue (General disorders) | 4 | 5
General physical health deterioration (General disorders) | 0 | 2
Influenza like illness (General disorders) | 1 | 1
Injection site pain (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 0 | 5
Pyrexia (General disorders) | 7 | 14
Hepatic pain (Hepatobiliary disorders) | 1 | 2
Cytokine release syndrome (Immune system disorders) | 1 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Lethargy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03256344/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03256344/SAP_001.pdf